CLINICAL TRIAL: NCT06023563
Title: Effect of Virtual Reality-based Training on Postural Control in Youth With Autism Spectrum Disorder
Brief Title: Effect of Virtual Reality-based Training on Balance and Walking in Youth With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Georgia Frey, Associate Professor, Public Health, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19116
Record Dates: First submitted 2023-07-17; First posted 2023-09-05 (Actual); Results first posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Balance exercises; Virtual reality; Active video gaming; Gait
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Two groups, intervention and the control, will be compared within and between longitudinally 3 times. Before-, after- and 4 weeks after the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Virtual reality active video gaming (Experimental): The participants in this group will engage in VR active gaming using Nintendo Switch Sports under supervision via Zoom, for 6 sessions over 2 weeks.
  Interventions: Device: Virtual reality active video gaming using Nintendo switch sports
- Standard balance exercises (Active Comparator): The participants in this group will engage in standard physical therapy exercises for balance and walking under supervision via Zoom, for 6 sessions over 2 weeks.
  Interventions: Behavioral: Standard physical therapy balance exercises

INTERVENTIONS:
Device: Virtual reality active video gaming using Nintendo switch sports — Playing 2 pre-selected VR active video games from beach tennis, soccer, volleyball, badminton, bowling, and chambara for 10 minutes each with a 5 minute break in-between. Total duration 30-40 minutes.
  Arms: Virtual reality active video gaming
Behavioral: Standard physical therapy balance exercises — Balance exercises: Standing with feet together for 10 seconds 5 times, standing with 1 foot in front of other for 10 seconds 5 times on both sides, standing on one leg for 10 seconds 5 times on both sides, walking with one foot in front of other on a 1-meter-long line for 5 repetitions and standing on a balance board for 30 seconds for 3 repetitions. 5 minutes each of warm-up and cool down exercises. Total duration 20-30 minutes.
  Arms: Standard balance exercises

SUMMARY:
The goal of this clinical trial is to assess the effect of short-term (3 days/week for 2 weeks) Virtual Reality (VR) active video gaming intervention on static and dynamic balance, versus traditional balance training exercises, in youth with ASD.

The participants in the intervention group will engage in VR active video gaming using the Nintendo Switch Sports under supervision via Zoom for 6 sessions occurring over 2 weeks, from their home. While, the participants in the control group will engage in standard physical therapy exercises for balance and walking under supervision via Zoom, for 6 sessions occurring over 2 weeks, from their home.

Their balance and walking will be assessed 3 times, 3-5 days before the intervention, 3-5 days after the intervention and 4-weeks after the intervention.

* Participants static balance will be assessed by standing on pressure mat, under 2 conditions, eyes open and eyes closed for 30 seconds each.
* The Pediatric Berg's balance Scale (PBS), a 14-point scale containing everyday activities, will be used as a clinical measure for assessing the static and dynamic balance.
* 13-infra-red camera motion capture system, Qualisys, will be used for assessing the walking.

The difference in the balance and walking parameters will be assessed and compared.

DETAILED DESCRIPTION:
Postural control deficits, also referred to as balance deficits, are a noted example of impaired motor-skills and are increasingly considered as one of the primary markers for autism spectrum disorder (ASD)1-5. However, there are very few controlled clinical trials examining effects of balance interventions in individuals with ASD. Moreover, to date there exist few effective interventions based on well-designed research that address balance deficits in youth with ASD and are home-implemented, cost-effective, generalizable, and enjoyable and that promote adherence. Virtual reality (VR) active gaming is one such intervention that incorporates scientific mechanisms for improving balance. But, there exist few, evidence-based best practices that use this method to address balance in youth with ASD. In addition to being based on principles of motor learning/control, commercially available VR active gaming can be affordable, enjoyable, at-home intervention. Thus, the aim of this study is to assess the effect of short-term (3 days/week for 2 weeks) Virtual Reality (VR) active video gaming intervention on static and dynamic balance, versus traditional balance training exercises, in youth with ASD.

This study will take place at the Physical Activity and Biomechanics Labs at School of Public Health, Indiana University, Bloomington, and participants home for total of 9 sessions occurring over 7-8 weeks.

Before participants come to the lab:

Participants' parent/guardian will complete a couple of questionnaires that will ask questions about any medications that participant takes and about participants' physical health to make sure it is safe for the participant to participate in the study. They will also answer questions that are used to determine if someone might have ASD.

Participants will be shown a video which will give them information about the lab they will be coming to do some of the study activities, and information about the people that will be working with them during the study. Participants will then be randomly assigned (like flipping a coin) to one of two groups: the Virtual Reality Group, or the Exercise Group. This will determine what activities or exercise they will do for the upcoming sessions.

Session #1, about 90 minutes:

Researchers measure participants height, weight, and length of arm and leg. Researchers will also measure which hand participants prefer to perform daily activities using Edinburgh Handedness Inventory- short form (EHI-SF). Participants will also stand on a large mat containing sensors that will measure how much their body moves back and forth while they are standing. Participants will stand on the mat for 30 seconds with their eyes open, and then for 30 seconds with their eyes closed.

Then, researchers will measure how well participants are able to balance by having them do some activities like sitting and standing without help, standing with their eyes closed, reaching forward with their arms stretched in front, placing their right then left foot on a stool, standing with alternating foot in front, and standing on one foot, alternating right and left. The researcher will show the participants how to do each of these, and they can practice a couple of times before the test begins.

Participants will then do some walking in the lab with special sensors that are attached to their lower back and feet. This will measure how participants walk. The sensors are attached with special tape to the cloths and shoes, and are not painful. A special camera will take pictures as the participants walk, and video recording will be done as well. Participants will do this several times and will be reminded to walk at a normal pace.

Lastly, if the participants are in the Virtual Reality Group, their parent/guardian will receive the Nintendo switch™ console and the sports game to take home.

At home, 3 times a week for two weeks for 30-40 minutes (Sessions 2-7):

* If participants are in the Virtual Reality Group, they will choose 2 video games on the Nintendo Switch from golf, Frisbee, beach tennis, soccer, Volleyball, badminton, bowling, and Chambara. Games will be played for 10 minutes each with a 5-minute break in-between. The same 2 games will be played at each session in the same sequence. Researchers will provide verbal prompts and encouragement during the games as they watch participants via Zoom. Each session will take approximately 30-40 minutes. Ideally, each session will occur with an off day in between, however this may not be realistic depending on participants schedules and so sessions will occur at their convenience.
* If participants are in the Exercise Group, they will perform balance exercises for 15 minutes with 5 minutes of warm and cool down each. Some of the exercises are standing with one foot in front of the other for 10 seconds, standing on 1 foot for 10 seconds, standing with feet together etc. Breaks will be given, and they will be given instructions and encouragement by the researcher who will be watching via Zoom.

Sessions 8 and 9 (in the lab), about an hour:

Session #8: 3-5 days after session 7, Participants will complete all the balance and walking measurements that they did in session #1 excluding parameters such as EHI-SF, leg and arm length, weight, height. It will take approximately 1 hour.

On session #9: 4 weeks after session #7, participants will once again complete all the same activities they completed during visit #8. It will take approximately 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* age 7-22 years,
* existing ASD DSM-5 level 1 or 2 diagnosis confirmed by medical record/ educational services categorized under ASD/ therapeutic services categorized under ASD/ any other official document indicating the diagnosis of ASD,
* able to follow instructions and
* able to stand unsupported for at least 20 minutes.

Exclusion Criteria:

* epilepsy or other medical conditions which can be exacerbated by looking at a screen,
* Uncorrected vision loss or any other eye condition prohibiting looking at the screen for a prolong time,
* co-occurring musculoskeletal conditions such as joint or muscle pain or stiffness that limits mobility, implanted plates, pins, or screws that limit mobility, fractures or recent surgeries or any other physical condition that could interfere with the ability to play an active video game
* co-occurring neurological conditions such as numbness or muscle weakness, temporary loss of vision, speech or strength, loss of consciousness (black out), Dizziness or lightheadedness, Impaired memory or confusion, any other cooccurring diagnosis that could be negatively impacted by playing an active video game
* any other health conditions that are contraindicated to or may interfere with physical activity such as impaired hearing (uncorrected), medically documented balance disorder, Any heart condition prohibiting exercise, chronic pain or any pain at the time of testing, need assistance to stand for 20 minutes or more,
* aggression or other severe behaviors that may limit the ability to safely participate in the intervention.

Ages: 7 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Georgia Frey, Ph.D., Principal Investigator — Indiana University, Bloomington
Locations (1):
- Indiana University Bloomington, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to maintain the confidentiality of the participants.

REFERENCES:
- [Background] Nobile M, Perego P, Piccinini L, Mani E, Rossi A, Bellina M, Molteni M. Further evidence of complex motor dysfunction in drug naive children with autism using automatic motion analysis of gait. Autism. 2011 May;15(3):263-83. doi: 10.1177/1362361309356929. Epub 2011 Apr 8. PMID 21478224
- [Background] Lim YH, Partridge K, Girdler S, Morris SL. Standing Postural Control in Individuals with Autism Spectrum Disorder: Systematic Review and Meta-analysis. J Autism Dev Disord. 2017 Jul;47(7):2238-2253. doi: 10.1007/s10803-017-3144-y. PMID 28508177
- [Background] Harris SR. Early motor delays as diagnostic clues in autism spectrum disorder. Eur J Pediatr. 2017 Sep;176(9):1259-1262. doi: 10.1007/s00431-017-2951-7. Epub 2017 Jun 28. PMID 28660313
- [Background] Li Y, Liu T, Venuti CE. Development of postural stability in children with autism spectrum disorder: a cross-sectional study. Int Biomech. 2021 Dec;8(1):54-62. doi: 10.1080/23335432.2021.1968316. PMID 34414860
- [Background] Minshew NJ, Sung K, Jones BL, Furman JM. Underdevelopment of the postural control system in autism. Neurology. 2004 Dec 14;63(11):2056-61. doi: 10.1212/01.wnl.0000145771.98657.62. PMID 15596750
- [Background] Mazurek MO, Shattuck PT, Wagner M, Cooper BP. Prevalence and correlates of screen-based media use among youths with autism spectrum disorders. J Autism Dev Disord. 2012 Aug;42(8):1757-67. doi: 10.1007/s10803-011-1413-8. PMID 22160370
- [Background] Ye S, Lee JE, Stodden DF, Gao Z. Impact of Exergaming on Children's Motor Skill Competence and Health-Related Fitness: A Quasi-Experimental Study. J Clin Med. 2018 Sep 7;7(9):261. doi: 10.3390/jcm7090261. PMID 30205483
- [Background] Bhat AN, Landa RJ, Galloway JC. Current perspectives on motor functioning in infants, children, and adults with autism spectrum disorders. Phys Ther. 2011 Jul;91(7):1116-29. doi: 10.2522/ptj.20100294. Epub 2011 May 5. PMID 21546566
- [Background] Ruggeri A, Dancel A, Johnson R, Sargent B. The effect of motor and physical activity intervention on motor outcomes of children with autism spectrum disorder: A systematic review. Autism. 2020 Apr;24(3):544-568. doi: 10.1177/1362361319885215. Epub 2019 Nov 29. PMID 31782658
- [Background] Zampella CJ, Wang LAL, Haley M, Hutchinson AG, de Marchena A. Motor Skill Differences in Autism Spectrum Disorder: a Clinically Focused Review. Curr Psychiatry Rep. 2021 Aug 13;23(10):64. doi: 10.1007/s11920-021-01280-6. PMID 34387753
- [Background] Jelsma D, Geuze RH, Mombarg R, Smits-Engelsman BC. The impact of Wii Fit intervention on dynamic balance control in children with probable Developmental Coordination Disorder and balance problems. Hum Mov Sci. 2014 Feb;33:404-18. doi: 10.1016/j.humov.2013.12.007. Epub 2014 Jan 18. PMID 24444657
- [Background] Rafiei Milajerdi H, Sheikh M, Najafabadi MG, Saghaei B, Naghdi N, Dewey D. The Effects of Physical Activity and Exergaming on Motor Skills and Executive Functions in Children with Autism Spectrum Disorder. Games Health J. 2021 Feb;10(1):33-42. doi: 10.1089/g4h.2019.0180. Epub 2020 Dec 23. PMID 33370161
- [Background] Travers BG, Mason AH, Mrotek LA, Ellertson A, Dean DC 3rd, Engel C, Gomez A, Dadalko OI, McLaughlin K. Biofeedback-Based, Videogame Balance Training in Autism. J Autism Dev Disord. 2018 Jan;48(1):163-175. doi: 10.1007/s10803-017-3310-2. PMID 28921103
- [Background] Caldani S, Atzori P, Peyre H, Delorme R, Bucci MP. Short rehabilitation training program may improve postural control in children with autism spectrum disorders: preliminary evidences. Sci Rep. 2020 May 13;10(1):7917. doi: 10.1038/s41598-020-64922-4. PMID 32404919
- [Background] Franjoine MR, Gunther JS, Taylor MJ. Pediatric balance scale: a modified version of the berg balance scale for the school-age child with mild to moderate motor impairment. Pediatr Phys Ther. 2003 Summer;15(2):114-28. doi: 10.1097/01.PEP.0000068117.48023.18. PMID 17057441
- [Background] Goetschius J, Feger MA, Hertel J, Hart JM. Validating Center-of-Pressure Balance Measurements Using the MatScan(R) Pressure Mat. J Sport Rehabil. 2018 Jan 1;27(1). doi: 10.1123/jsr.2017-0152. Epub 2018 Jan 24. PMID 28714837
- [Background] Chen CL, Shen IH, Chen CY, Wu CY, Liu WY, Chung CY. Validity, responsiveness, minimal detectable change, and minimal clinically important change of Pediatric Balance Scale in children with cerebral palsy. Res Dev Disabil. 2013 Mar;34(3):916-22. doi: 10.1016/j.ridd.2012.11.006. Epub 2013 Jan 3. PMID 23291508

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Virtual Reality Active Video Gaming | Standard Balance Exercises
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Virtual Reality Active Video Gaming | Standard Balance Exercises | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 4
  Between 18 and 65 years | 5 | 4 | 9
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.14 (5.49) | 16.0 (6.03) | 17.0 (5.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 5 | 5 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change in the Center of Pressure Movement (Postural Sway Velocity)
Description: High resolution pressure mat containing multiple integrated sensors is used to detect center of pressure movement of the person standing on it recorded at 100 Hz
Time Frame: 5 days before the intervention, 5 days after the intervention and 4 weeks after the intervention
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | Virtual Reality Active Video Gaming | Standard Balance Exercises
Number analyzed (Participants) | 7 | 6
cm/sec
  baseline | 0.93 (1.02) | 0.50 (0.30)
  post-1 | 1 (1.1) | 0.8 (0.69)
  post-2 | 1.4 (2.1) | 0.74 (0.63)
Statistical Analysis 1: Comparison: Virtual Reality Active Video Gaming vs Standard Balance Exercises; A virtual reality active video gaming intervention will be more effective than traditional physical therapy based balance exercises, both based on motor learning principles, in improving static and dynamic balance in youth and young adults with ASD and these improvements will be retained at 4 weeks after the intervention; Test type: Other — The required sample size for medium effect size (f = 0.25) and power of 0.80 was calculated to be 6 participants in each group (n =12) (G*power 3.1.9.7 software). Data were analyzed using IBM SPSS statistical package (version 29.0.1.0); p < 0.05, Friedman's test

2. Primary Outcome: Change in Pediatric Berg's Balance Scale Score
Description: Pediatric Berg's balance Scale: 14-component battery that evaluates daily living tasks such as sitting to standing, transferring from one chair to another, and sitting and standing without support. This scale is reliable and valid clinical balance assessment tool for children and youth with motor impairments. Maximum total score is 56 points and minimum total score is 0 points. Higher score indicates better balance such that increase in total score by 3.7 points indicates minimal clinically important difference.
Time Frame: 5 days before the intervention, 5 days after the intervention, 4 weeks after the intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality Active Video Gaming | Standard Balance Exercises
Number analyzed (Participants) | 7 | 6
score on a scale
  baseline | 51.86 (2.91) | 52.00 (2.00)
  post-1 | 55.43 (1.13) | 55 (1.26)
  post-2 | 55.14 (1.21) | 54.67 (1.21)
Statistical Analysis 1: Comparison: Virtual Reality Active Video Gaming vs Standard Balance Exercises; Test type: Other; p < 0.05, Friedman's test

3. Primary Outcome: Change in Step Length (Meters) of the Gait
Description: 13-infra red camera system with 19-light reflecting passive markers recording at 100 Hz are used to measure the gait parameter: step length (meters).
Time Frame: 5 days before the intervention, 5 days after the intervention, 4 weeks after the intervention
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Virtual Reality Active Video Gaming | Standard Balance Exercises
Number analyzed (Participants) | 7 | 6
m
  Baseline | 0.69 (0.07) | 0.71 (0.03)
  post-1 | 0.68 (0.12) | 0.66 (0.06)
  post-2 | 0.71 (0.06) | 0.70 (0.07)
Statistical Analysis 1: Comparison: Virtual Reality Active Video Gaming vs Standard Balance Exercises; Test type: Other; p < 0.05, Friedman's test

4. Primary Outcome: Change in Stride Width (Meters) of the Gait
Description: 13-infra red camera system with 19-light reflecting passive markers recording at 100 Hz are used to measure the gait parameter: step width (meters).
Time Frame: 5 days before the intervention, 5 days after the intervention, 4 weeks after the intervention
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Virtual Reality Active Video Gaming | Standard Balance Exercises
Number analyzed (Participants) | 7 | 6
m
  Baseline | 0.11 (0.03) | 0.11 (0.03)
  post-1 | 0.11 (0.03) | 0.11 (0.02)
  post-2 | 0.12 (0.03) | 0.11 (0.02)
Statistical Analysis 1: Comparison: Virtual Reality Active Video Gaming vs Standard Balance Exercises; Test type: Other; p < 0.05, Friedman's test

5. Primary Outcome: Change in Stride Length (Meters) of the Gait
Description: 13-infra red camera system with 19-light reflecting passive markers recording at 100 Hz are used to measure the gait parameter: stride length (meters).
Time Frame: 5 days before the intervention, 5 days after the intervention, 4 weeks after the intervention
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Virtual Reality Active Video Gaming | Standard Balance Exercises
Number analyzed (Participants) | 7 | 6
m
  Baseline | 1.33 (0.14) | 1.37 (0.05)
  post-1 | 1.35 (0.14) | 1.31 (0.15)
  post-2 | 1.37 (0.14) | 1.38 (0.14)
Statistical Analysis 1: Comparison: Virtual Reality Active Video Gaming vs Standard Balance Exercises; Test type: Other; p < 0.05, Friedman's test

6. Primary Outcome: Change in Double Support Period (Seconds) of the Gait
Description: 13-infra red camera system with 19-light reflecting passive markers recording at 100 Hz are used to measure the gait parameter: double support period (seconds).
Time Frame: 5 days before the intervention, 5 days after the intervention, 4 weeks after the intervention
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Virtual Reality Active Video Gaming | Standard Balance Exercises
Number analyzed (Participants) | 7 | 6
sec
  Baseline | 0.12 (0.03) | 0.15 (0.03)
  post-1 | 0.11 (0.02) | 0.17 (0.05)
  post-2 | 0.12 (0.04) | 0.15 (0.03)
Statistical Analysis 1: Comparison: Virtual Reality Active Video Gaming vs Standard Balance Exercises; Test type: Other; p < 0.05, Friedman's test

7. Primary Outcome: Change in the Cadence (Steps/Minute) of the Gait
Description: 13-infra red camera system with 19-light reflecting passive markers recording at 100 Hz are used to measure the gait parameter: cadence (number of steps/minute).
Time Frame: 5 days before the intervention, 5 days after the intervention, 4 weeks after the intervention
Measure: Mean (Standard Deviation); unit: steps/min
Arm/Group | Virtual Reality Active Video Gaming | Standard Balance Exercises
Number analyzed (Participants) | 7 | 6
steps/min
  baseline | 111.96 (9.89) | 110.31 (4.85)
  post-1 | 114.70 (8.98) | 115.80 (14.97)
  post-2 | 113.76 (6.52) | 113.71 (3.51)
Statistical Analysis 1: Comparison: Virtual Reality Active Video Gaming vs Standard Balance Exercises; Test type: Other; p < 0.05, Friedman's test

8. Primary Outcome: Change in Gait Velocity (Meters/Second)
Description: 13-infra red camera system with 19-light reflecting passive markers recording at 100 Hz are used to measure the gait parameter: gait velocity (meters/second).
Time Frame: 5 days before the intervention, 5 days after the intervention, 4 weeks after the intervention
Measure: Mean (Standard Deviation); unit: m/sec
Arm/Group | Virtual Reality Active Video Gaming | Standard Balance Exercises
Number analyzed (Participants) | 7 | 6
m/sec
  baseline | 1.27 (0.21) | 1.25 (0.10)
  post-1 | 1.30 (0.20) | 1.20 (0.12)
  post-2 | 1.30 (0.18) | 1.29 (0.09)
Statistical Analysis 1: Comparison: Virtual Reality Active Video Gaming vs Standard Balance Exercises; Test type: Other; p < 0.05, Friedman's test

ADVERSE EVENTS:
Time Frame: 44 weeks
Description: The participants were not at a risk of acquiring/ experiencing adverse events or mortality risk as it is a behavioral intervention, comparing two methods of administrating physical therapy for improving static and dynamic balance in youth and young adults with ASD. Minimal fall risk was mitigated through presence of chair at a hands distance from participants to grab in destabilizing condition and presence of caregiver in the room for entirety of intervention sessions.
Arm/Group | Virtual Reality Active Video Gaming | Standard Balance Exercises
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/6

LIMITATIONS AND CAVEATS:
Limitations:

Both interventions were carried out under video supervision, and this may have impacted motivation.

All balance data was collected in laboratory-based setting. Findings therefore may not be generalizable to postural balance mechanics during outdoor or free-living walking.

Gender-based differences were present in the sample as prevalence of ASD is 4:1 male to female ratio

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-01-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT06023563/Prot_SAP_ICF_001.pdf